CLINICAL TRIAL: NCT00001325
Title: Natural History of Metabolic Abnormalities in Children With Epilepsy
Brief Title: Metabolic Abnormalities in Children With Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920175; 92-N-0175
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-06

CONDITIONS: Generalized Epilepsy; Infantile Spasms; Metabolic Disease; Partial Epilepsy; Seizures
Keywords: Positron; Tomography; Seizures; Epileptic Focus; Electroencephalography; Metabolism; Glucose; Cerebral; Positron Emission Tomography; Lennox Gastaut Syndrome
MeSH Terms: conditions — Epilepsy, Generalized; Spasms, Infantile; Metabolic Diseases; Epilepsies, Partial; Seizures; Lennox Gastaut Syndrome | interventions — Fluorodeoxyglucose F18

INTERVENTIONS:
Drug: 18 FDG

SUMMARY:
This study is designed to use positron emission tomography to measure brain energy use. Positron Emission Tomography (PET) is a technique used to investigate the functional activity of the brain. The PET technique allows doctors to study the normal processes of the brain (central nervous system) of normal individuals and patients with neurologic illnesses without physical / structural damage to the brain.

When a region of the brain is active, it uses more fuel in the form of oxygen and sugar (glucose). As the brain uses more fuel it produces more waste products, carbon dioxide and water. Blood carries fuel to the brain and waste products away from the brain. As brain activity increases blood flow to and from the area of activity increases also.

Researchers can label a sugar with a small radioactive molecule called FDG (fluorodeoxyglucose). As areas of the brain use more sugar the PET scan will detect the FDG and show the areas of the brain that are active. By using this technique researchers hope to answer the following questions;

4. Are changes in brain energy use (metabolism) present early in the course of epilepsy

5. Do changes in brain metabolism match the severity of patient's seizures

6. Do changes in metabolism occur over time or in response to drug therapy

DETAILED DESCRIPTION:
We propose to study children with recent onset partial epilepsy, cryptogenic infantile spasms, and idiopathic Lennox-Gastaut Syndrome with serial FDG-PET to elucidate the natural history and evolution of metabolic abnormalities associated with such epilepsies. The severity of the seizure disorder, and cognitive impairment, when present, will be correlated with the presence and extent of focal and global cerebral metabolic abnormalities.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with partial seizures, infantile spasms and Lennox-Gastaut syndrome will be selected.

EXCLUSION CRITERIA:

Evidence of a structural lesion as cause for epilepsy.

Degenerative or metabolic disease.

Inability to comply with the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 1992-04; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bourgeois BF, Prensky AL, Palkes HS, Talent BK, Busch SG. Intelligence in epilepsy: a prospective study in children. Ann Neurol. 1983 Oct;14(4):438-44. doi: 10.1002/ana.410140407. PMID 6416142
- [Background] Chugani HT, Phelps ME, Mazziotta JC. Positron emission tomography study of human brain functional development. Ann Neurol. 1987 Oct;22(4):487-97. doi: 10.1002/ana.410220408. PMID 3501693
- [Background] Engel J Jr, Kuhl DE, Phelps ME, Mazziotta JC. Interictal cerebral glucose metabolism in partial epilepsy and its relation to EEG changes. Ann Neurol. 1982 Dec;12(6):510-7. doi: 10.1002/ana.410120603. PMID 6818896